CLINICAL TRIAL: NCT04766255
Title: Behavioral Comparison of Three Different Graft Materials to Increase Soft Tissue Thickness Around Dental Implants in Terms of Volume Gain and Stability Over Time: A Randomized Clinical Trial.
Brief Title: Behavioral Comparison of Three Different Graft Materials to Increase Soft Tissue Thickness Around Dental Implants.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Andres Pascual La Rocca, Master in Periodontics program director, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PER-ECL-2017-07
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Soft Tissue Atrophy; Mucogingival Deformity on Edentulous Ridge; Edentulous Alveolar Ridge
Keywords: soft tissue graft; acellular dermal graft; collagen matrix

STUDY DESIGN:
Intervention Model Description: controlled randomized prospective clinical study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Control Group (Active Comparator): Implant placement and prosthetic rehabilitation of the missing tooth
  Interventions: Procedure: Implant Placement
- SCTG group (Experimental): Implant placement, soft tissue augumentation of Connective Tissue Graft (from the palate) (SCTG) at the implant site and prosthetic rehabilitation of the missing tooth.
  Interventions: Procedure: Soft Tissue graft augmentation; Procedure: Implant Placement
- CM group (Experimental): Implant placement, soft tissue augumentation of porcine collagen matrix (CM) at the implant site and prosthetic rehabilitation of the missing tooth.
  Interventions: Procedure: Soft Tissue graft augmentation; Procedure: Implant Placement
- PADM group (Experimental): Implant placement, soft tissue augumentation of Porcine acellular dermal matrix (PADM) at the implant site and prosthetic rehabilitation of the missing tooth.
  Interventions: Procedure: Soft Tissue graft augmentation; Procedure: Implant Placement

INTERVENTIONS:
Procedure: Soft Tissue graft augmentation — Donor site:
  SCTG group: The SCTG will be harvested in the palat,In order to extract the same thickness in each grafts a double-bladed knife (separated by 1,5mm) will be used. The donor area will be sutured.
  Recipient site:
  SCTG group: the connective tissue graft will be trimmed to the correct dimensions (10mm height, 12mm length and 1,5mm thick) and placed and secured at the recipient site with a resorbable 5-0 suture CM group: The CM graft (Geistlich Fibro-gide) will be trimmed to the indicated dimensions (10mm height, 12mm length) and placed and secured at the recipient site with resorbable 5-0 suture PADM Group: the ADM (NovoMatrix, Biohorizons, Birmingham AL) graft will be trimmed to the indicated dimensions (10mm height, 12mm length) and placed and secured at the recipient site with resorbable 5-0 suture
  Arms: CM group; PADM group; SCTG group
Procedure: Implant Placement — A crestal incision will be made in the implant reception area, extending from the distal of the most mesial tooth to the mesial of the most distal tooth. A mucoperiosteal flap will be elevated in the most crestal part of the ridge. The receptor bed will be prepared following the established drilling protocol for the placement of a BioHorizons Tapered Pro Implant (Biohorizons, Birmingham AL). The diameter and length of the implant will be previously established during the implant study. Later a healing abutment will be placed.

SUMMARY:
The purpose of the study is to compare soft tissue volume changes in terms of volume gain and stability around dental implants and PROMS in cases where a sub-epithelial connective tissue graft (SCTG) from the palate, Porcine collagen matrix (CM) or Porcine Acellular dermal matrix (PADM) is used after 3 and 15 months after implant placement.

ELIGIBILITY:
Inclusion Criteria:

Patients referred to Department of Periodontology (CUO) in need of a single implant and need of soft tissue augmentation such as buccal defects, thin biotype, lack of keratinized tissue and aesthetic compromised situation.

* The patient must be ≥18 years and able to understand the nature of the proposed surgery and must sign an informed consent.
* The implant must be located between 2 fixed reference points (i.e. clinical crowns).
* Anterior and premolar teeth (from premolar to premolar).
* Enough crestal bone width to leave a minimum thickness of 2mm at the buccal bone plate when placing the implant.
* Palate must have ≥2mm of thickness at premolar area.
* Full mouth plaque and bleeding score <20%.

Exclusion Criteria:

* Pregnant or lactation.
* Active periodontal disease.
* Previous soft tissue augmentation in the area.
* Need of guided bone regeneration (GBR) during or after the placement of the implant.
* Heavy smokers (> 10 cigarettes per day).
* Local or systemic conditions that would interfere with routine periodontal therapy (non-controlled diabetes mellitus, cancer, HIV, Chronic High dose steroid therapy, bone metabolic diseases, radiation, immunosuppressive disorders, liver function disorder, immunosuppressant disease, autoimmune disease).
* Allergy to non-steroidal anti-inflammatory drugs.
* Patients taking medications that cause gingival enlargement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
soft tissue volume gain | after 3 months
  Optical scans superposition

SECONDARY OUTCOMES:
soft tissue volume stability | after 15 months
  Optical scans superposition
Plaque index (PI) | at baseline, after 12 weeks and after 15 months.
  Each tooth will be divided in 4 surfaces: buccal, lingual, mesial, distal. After the application of erythrosine, O'Leary plaque index will be registered (O'Leary et al. 1972)
Bleeding on probing (BI) | at baseline, after 12 weeks and after 15 months.
  Each tooth will be divided in 4 surfaces: buccal, lingual, mesial, distal. After a gentle probing if the gingiva bleeds will be positive.
Probing depth (PD) | at baseline, after 12 weeks and after 15 months.
  in the implant area (implant and both tooth next to it). Distance from the gingival margin to the bottom of the gingival sulcus using periodontal probe (UNC 15). Measured in 6 points: mesiobuccal, buccal, distobuccal, mesiolingual, lingual and distolingual.
Width of keratinized tissue (KT) | at baseline, after 12 weeks and after 15 months.
  in the implant area (implant and both teeth nxt to it). Measured in the medial buccal point of the tooth/implant. Distance from mucogingival junction to the most apical portion of the crest of the marginal gingiva. The mucogingival junction will be identified by the roll technique, wherein the mucosa is rolled until the non-movable portion of the attached keratinized tissue is seen
Phenotype evaluation (PT) | at baseline, after 12 weeks and after 15 months.
  the gingival biotype was categorized as thin or thick based on the transparency of a periodontal probe (CP15 UNC; Hu-Friedy, Chicago, IL, USA) through the soft tissues while probing the buccal sulcus of the contra-lateral tooth (17-19)
Patient reported outcome measures (PROMs) | after the surgery procedures (baseline) and after 7 days (suture removal)
  patient pain/discomfort will be evaluated (a questionnaire will be provided to each patient after all the surgery procedures and it will be recollected the day of suture removal)
Pink Esthetic Score (PES) | After 2 weeks of the definite crown placement (around 16 months)
  will be registered to obtain information related to the papilla, the level of soft-tissue margin, the alveolar process, the color, contour and texture of the same soft tissue

CONTACTS AND LOCATIONS:
Overall Officials: Andres Pascual La Rocca, DDS, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No